CLINICAL TRIAL: NCT05007574
Title: A Prospective Observational Pilot Study to Evaluate the Reliability and Usability of a Microphone Connected to a Medical Data Analysis Platform to Monitor Coughs in Hospitalized Patients Suffering From Respiratory Diseases
Brief Title: A Microphone for Monitoring Coughs
Acronym: CoughMonit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ligue Pulmonaire Neuchâteloise (Other)
Responsible Party: Sponsor
Other Study IDs: LPNE_03
Record Dates: First submitted 2021-07-07; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Disease
Keywords: cough; exacerbation; connected device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiration Disorders; Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Microphone MI-305 — Remote data collection

SUMMARY:
Aging of the population is dramatically increasing the number of hospitalized patients, with the consequent challenges of limited medical personnel and resources in hospitals. Wireless technologies that create highly connected healthcare environments are developed to help hospitals address these issues, once these technologies are perfectly integrated in the hospital environment with respect to IT infrastructure for big data storage. Such devices have proven remarkable efficiencies in monitoring patients with high patient safety, data accuracy and security, which are essential to provide high quality patient care, reduce health-related costs and optimize the management of high numbers of patients.

Cough is the most common condition that results in a visit to the physician. Often coughs are benign, but sometimes can be the sign of exacerbations of a chronic respiratory disease. Exacerbations are defined in the Global Initiative for Chronic Obstructive Lung Disease (GOLD) document "as an acute event characterised by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication". It is assumed that, if coughs were remotely monitored, hospitals might be unburdened, patients would be empowered to self-manage their health, and that prevention of serious respiratory diseases might be facilitated, thus improving health outcomes. Unfortunately, remote monitoring for cough that rely on self-reporting is impractical, as patients do not record data very reliably. On the contrary, a microphone on the bedside table connected to a medical data analysis platform might monitor patients' cough exacerbations at night and alert the medical staff immediately.

DETAILED DESCRIPTION:
The clinical study is designed as a prospective observational pilot study to evaluate the reliability of a microphone and data analysis platform to monitor coughs in hospitalized patients with respiratory diseases.

The study includes three phases:

1. Calibration phase: to determine the degree of coughs' homogeneity between patients. The control source of data will be a polygraph to record cough events and movements. Polygraphy is the conventional method currently used to analyse night coughing.

   At the end of the calibration period, the data generated by the device will be analysed to determine if the coughs are homogeneous or heterogeneous, according to patient follow-up and polygragh outcomes. The degree of homogeneity will allow establishing the correct number of patients to be followed in the interventional phase (estimated 20 patients) and to set a threshold to define when there is an exacerbation.
2. Observational phase: to collect data in about 20 patients from sources, namely the microphone and the polygraph in the patient's room. Data will be collected in parallel by the two systems during two consecutive nights for each patient.
3. Data analysis phase: to correlate microphone and polygraph signals. These results will be reported in a format provided by the device supplier. Subsequently, specialized engineers will correlate the polygraph results with the microphone's signals. .

ELIGIBILITY:
Inclusion Criteria:

* Suffering from chronic obstructive pulmonary disease (COPD I to IV) or other respiratory diseases generating dry or productive cough and hospitalized for a minimal duration of 5 days
* Living in the Canton of Neuchâtel
* Understanding French

Exclusion Criteria:

* Suffering from cognitive disorders
* Refractory to test new technologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects aged ≥ 18 years fulfilling all of the inclusion criteria are eligible for the study. The presence of any one of the exclusion criteria will lead to exclusion of the participant.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the clinical performance and accuracy of the microphone and of the analysis platform to detect coughs | 2 nights
  The microphone signal is recorded by a micro-computer and treated by the algorithm of the analysis platform developped by the company VNV. The aim of this algorithm is to discriminate events of cough in the signal.
  To measure the accuracy of the algorithm, we will compare the results obtained by the analysis plateform with a polygraph which is the classical way to measure night cough. The microphone of the polygraph placed on the patient chest will control if the events are due to patients coughs or patient movements.
  The 2 devices (microphone and polygraph) will be recording patients during 2 consecutive nights.
  Unit of measurement will be the number of cough events.

SECONDARY OUTCOMES:
Patients' acceptance on the connected microphone | 2 nights
  Determination of the level of acceptance of the microphone by patients by means of a patient questionnaire to provide feedback. Usability for patients will be assessed by the % rate of acceptance for the patients. This questionnaire has been developped by the pneumology service of Hôpital Neuchâtelois.
  The different items to rate/answer are:
  * Clarity of informations about the device
  * Reason of the study participation
  * Ease of use
  * Suggestions or complaints
Medical staff's satisfaction on both the microphone and the medical analysis platform (usability, data usage) | 5 days
  Assessment of the satisfaction of the medical staff regarding the usability of the microphone and of the microphone-generated data by means of a health professional questionnaire to provide feedback. Usability for healthcare professionals will be assessed by the % rate of satisfaction for the healthcare professionals.
  This questionnaire has been developped by the pneumology service of Hôpital Neuchâtelois.
  The different items to rate/answer are:
  * Installation of the device
  * Training on the use of the device
  * Ease of use
  * Advantages and disadvantages
  * Compatibility of the device on patients with respiratory diseases
  * Usefulness
  * Recommandation of the device to other health professionnels
  * Use of the device at the hospital
  * Use of the device at home
  * Suggestions

CONTACTS AND LOCATIONS:
Locations (1):
- Ligue pulmonaire neuchâteloise, Peseux, Canton of Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided